CLINICAL TRIAL: NCT05476224
Title: Qualitative and Functional Investigation of Lipids in Patients With SARS-CoV2 Infection - In Search of Atherogenic Sequelae
Acronym: COVI-LIPI-D
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ROULAND ANRS 2022
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A history of asymptomatic/mildly symptomatic SARS-CoV2 infection: Participant with asymptomatic or mild symptomatic SARS CoV2 infection that did not require hospitalization at least 6 months prior to study inclusion
  Interventions: Biological: Blood sample of 30 ml
- A history of symptomatic SARS-CoV2 infection hospitalized at the CHU of Dijon outside the ICU: participant with symptomatic SARS CoV2 infection requiring conventional hospitalization at least 6 months prior to study inclusion
  Interventions: Biological: Blood sample of 30 ml
- A history of symptomatic SARS-CoV2 infection hospitalized in the ICU: participant with a symptomatic SARS CoV2 infection requiring an ICU hospitalization at least 6 months prior to study inclusion
  Interventions: Biological: Blood sample of 30 ml
- No history of SARS-CoV2 infection matched on sex and age: participant with no evidence of SARS CoV2 infection and negative SARS-CoV2 serology
  Interventions: Biological: Blood sample of 30 ml

INTERVENTIONS:
Biological: Blood sample of 30 ml — The parameters analyzed on this blood sample: Fasting blood glucose, HbA1C, creatinine, creatinine clearance (MDRD), fasting lipid profile (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides.

SUMMARY:
Currently, the world is facing a SARS-CoV2 coronavirus epidemic, which is responsible for COVID-19. In France, this virus has already infected several million people and is responsible for the death of more than 127,000.

Infection is associated with a higher number of cardiovascular events (myocardial infarction, stroke, cardiac arrhythmia, thrombosis ...) in the short and medium term after infection. The long-term complications of this infection are not yet known and are the subject of research in France and in the world.

In order to investigate the possible long term sequelae of this virus infection, this research aims to evaluate the potential cholesterol abnormalities caused by COVID-19, which could play a significant role in the increase of cardiovascular risk in affected patients.

A total of 180 analysable participants will be recruited in this study. They will be divided into four groups of participants that will be compared to one another:

* 30 participants who were infected with SARS-CoV2 with no or few signs and did not require hospitalization.
* 30 participants who were infected with SARS-CoV2 and whose severity of illness required hospitalization in a COVID unit
* 30 participants who were infected with SARS-CoV2 and required intensive care hospitalization due to severity of illness.
* 90 participants who were not infected with SARS-CoV2.

For each participant, the study will last approximately 1 hour, the time to fill out the consent forms, to answer a few questions about their current medical history and finally to take a blood sample for lipid measurements.

ELIGIBILITY:
Inclusion Criteria:

Participants with a history of asymptomatic/mildly symptomatic SARS-CoV2 infection:

* Age ≥18 years
* Participant who has provided consent
* Participant affiliated to National health insurance
* Participant with asymptomatic or minimally symptomatic SARS CoV2 infection who did not require hospitalization at least 6 months prior to study inclusion.
* SARS CoV2 infection proven by positive PCR or antigenic test at the time of signs of infection or positive SARS-CoV2 infection-specific serology at the time of infection (IgG+).

Participants with a history of symptomatic SARS-CoV2 infection hospitalized at the Dijon University Hospital excluding the intensive care unit:

* Age ≥18 years
* Participant having provided consent
* Participant affiliated to National health insurance
* Participant having presented a symptomatic SARS CoV2 infection requiring admission to a regular hospital unit at least 6 months prior to inclusion in the study.
* SARS CoV2 infection proven by a positive PCR or antigenic test at the time of signs of infection or a positive SARS-CoV2 specific serology at the time of infection (IgG+).

Participants with a history of symptomatic SARS-CoV2 infection hospitalized at Dijon University Hospital in the ICU:

* Age ≥18 years
* Participant who has provided consent
* Participant affiliated to National health insurance
* Participant with symptomatic SARS CoV2 infection requiring admission to an intensive care unit at least 6 months prior to study inclusion.
* SARS CoV2 infection proven by a positive PCR or antigenic test at the time of signs of infection or a positive SARS-CoV2 specific serology at the time of infection (IgG+).

Participants with no history of SARS-CoV2 infection:

* Age≥18 years
* Participant who has provided consent
* Participant affiliated to National health insurance
* Participant with no evidence of SARS CoV2 infection and negative SARS-CoV2 serology.
* For vaccinated participants: negative specific serology for SARS-CoV2 infection

Exclusion Criteria:

For all participants:

* SARS Cov2 vaccination within one month prior to inclusion.
* Previous SARS Cov1 infection documented
* Previous study participant
* Participant under legal protection (guardianship)
* Participant subject to a legal protection measure
* A protected adult
* Pregnant, parturient or breastfeeding women
* Treatment with corticosteroids in the last year
* Treatment with lipid-lowering drugs
* Known genetic mutation modifying HDL cholesterol
* Progressive neoplasia
* Chronic alcoholism
* Primary biliary cirrhosis
* Hyperthyroidism
* Unstable hypothyroidism
* History of cardiac or cardiovascular side effects following SARS-CoV2 vaccination (thrombosis, myocarditis etc)

For participants with a history of asymptomatic/mildly symptomatic SARS-CoV2 infection:

- Hospitalization with a prior SARS-CoV2 infection in a conventional or intensive care unit

For participants with a history of symptomatic SARS-CoV2 infection hospitalized outside the ICU:

- Previous ICU hospitalization for SARS-CoV2 infection

For participants with no history of SARS-CoV2 infection:

* Previous positive SARS-CoV2 PCR
* Negative SARS-CoV2 PCR and presence of clinical symptoms suggestive of SARS-CoV2 infection
* Previous positive serology for SARS-CoV2 infection

Secondary exclusion criteria :

For healthy volunteers with no history of SARS-CoV2 infection:

Positive specific serology for SARS-CoV2 infection at the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SARS-CoV2 infection
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration expressed as a percentage of sphingomyelin to total HDL mass | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France